CLINICAL TRIAL: NCT06870903
Title: Comparison of Transvaginal Paracervical and Transperitoneal Approaches in Lymphadenectomy During v-NOTES Surgery for Patients Diagnosed With Endometrial Cancer
Acronym: ENDONOTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sedat Akgöl, Head of Gynecology Oncology Department, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENDOCA
Record Dates: First submitted 2025-02-25; First posted 2025-03-11 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Endometrial Cancer; Lymphadenectomy; Sentinel Lymph Node Biopsy; Minimally Invasive Surgical Procedures; Natural Orifice Transluminal Endoscopic Surgery
Keywords: endometrial cancer; V-NOTES; lymphadenectomy; sentinel lymph node; transperitoneal; extraperitoneal
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transvaginal paracervical sentinel lymphadenectomy group (Experimental): Surgical Procedure of transvaginal sentinel lymphadenectomy group:
  All patients will be operated in accordance with Memorial Sloan Kettering Cancer Center procedure. V-NOTES will consist of transvaginal paracervical sentinel lymph node (SLN) mapping followed by V-NOTES hysterectomy and bilateral salpingo-oophorectomy (BSO).
  SLN Mapping:
  Under general anesthesia, subjects will be placed in supine lithotomy position. Methylene blue solution (BLUMET IV INJECTION INJECTABLE 50 mg/5 ml 1x5 ml) (1 mL submucosal to the cervix at the 3 and 9 o'clock positions and 1 mL at a depth of 1-2 cm, using a total volume of 2-4 mL.
  Monitoring of lymphatic ducts includes identification of structures stained with methylene blue dye in the expected anatomical location, typically between the internal and external iliac veins or in the obturator region. Bilateral and symmetrical structures believed to be sentinel lymph nodes (SLNs) will be removed. When unilate
  Interventions: Procedure: Extraperitoneal(transvaginal paracervical sentinel lymphadenectomy) group lymphadenectomy
- Transperitoneal lymphadenectomy (Active Comparator): In this arm, patients will undergo transperitoneal lymphadenectomy with V-NOTES. The procedure begins with methylene blue injection for sentinel lymph nodes. Methylene blue will be injected at the 3 and 9 o'clock positions on the cervix, first at a depth of 1 mm and then at 4 mm, with 1 cc administered at each point. This will result in a total of 4 cc (1 cc x 4). Then, the procedure will continue with anterior and posterior colpotomies, followed by placement of the V-NOTES apparatus. Hysterectomy is performed first, followed by peritoneal dissection and lymph node excision.
  Interventions: Procedure: Transperitoneal lymphadenectomy

INTERVENTIONS:
Procedure: Extraperitoneal(transvaginal paracervical sentinel lymphadenectomy) group lymphadenectomy — The procedure begins with a vaginal incision in the lateral vaginal fornices (on both sides), which is then extended to allow placement of the V-NOTES apparatus. By identifying an appropriate cleavage plane, the obturator fossa is accessed to excise the obturator lymph nodes. Following this, an anterior colpotomy is performed to access the vesicocervical space, and a posterior colpotomy is made to open the rectouterine pouch. The V-NOTES apparatus is then placed to continue with the hysterectomy and bilateral salpingo-oophorectomy (BSO).
  Arms: transvaginal paracervical sentinel lymphadenectomy group
Procedure: Transperitoneal lymphadenectomy — In this arm, patients will undergo transperitoneal lymphadenectomy with V-NOTES. The procedure begins with anterior and posterior colpotomies, followed by placement of the V-NOTES apparatus. Hysterectomy is performed first, followed by peritoneal dissection and lymph node excision.
  Arms: Transperitoneal lymphadenectomy

SUMMARY:
The aim of this study is to compare two types of lymphadenectomy (transperitoneal vs. paracervical) during the lymphadenectomy phase of endometrial cancer staging surgery performed using V-NOTES, a new and advanced technique. This study seeks to optimize the V-NOTES technique for endometrial cancer staging. This randomized, prospective, controlled study will include patients diagnosed with endometrial cancer via histology, following physical examination and imaging, and who are electively scheduled for the V-NOTES endometrial cancer staging procedure. Patients will be randomized into two groups: the transvaginal paracervical lymphadenectomy group and the transperitoneal lymphadenectomy group. The parameters related with surgical and functional outcomes will be compared in both groups.

DETAILED DESCRIPTION:
Surgical staging is often the primary management strategy for endometrial cancer. Sentinel lymph node (SLN) procedures are considered an alternative standard of care in the treatment of significant uterus-confined malignancy. Both accurately estimate nodal status and reduce the surgical morbidity associated with complete lymphadenectomy. Laparoscopic surgery for endometrial cancer has been associated with equal or better quality of life, less blood loss and similar cancer-related outcomes. A new innovation, natural orifice transluminal endoscopic surgery (NOTES), has been developed to further reduce morbidity and scarring associated with laparoscopic surgery. NOTES utilizes the natural orifices of the human body for access to the peritoneal cavity when performing endoscopic surgery.

However, there is no standardization in vNOTES SLN mapping and lymph tracers are diverse. Many procedures and tracers have been reported, such as intra- or retroperitoneal surgery, a range of vaginal surgeries, SLN exposure method, and indocyanine green or methylene blue injection, and they lack comparative studies. This study will evaluate feasibility and surgical outcomes by comparing transvaginal paracervical and transperitoneal mapping in vNOTES hysterectomy with SLN procedure in endometrial cancer.

The study is an observational study with a prospective design. It will be implemented in a single institution, specifically Diyarbakır Gazi Yaşargil Training and Research Hospital, which functions as a tertiary cancer treatment facility.

Between March 2025 and December 2025, patients with newly diagnosed clinical early stage (FIGO 2023 stages 1 and 2) endometrial cancer who will be treated with laparoscopic surgical staging with SLN mapping.

According to inclusion and exclusion criteria, the patients will be randomized into two groups: the transvaginal paracervical lymphadenectomy group and the transperitoneal lymphadenectomy group.

Surgical Procedure of transvaginal paracervical sentinel lymphadenectomy group:

All patients(26) will receive V-NOTES with transvaginal paracervical sentinel lymph node (SLN) mapping followed by V-NOTES hysterectomy and bilateral salpingo-oophorectomy (BSO).

Transperitoneal sentinel lenfadenectomy group's Surgical Procedure:

All patients (26) will receive vNOTES hysterectomy with bilateral salpingo-oophorectomy (BSO) followed by transperitoneal vNOTES sentinel lymph node (SLN) mapping.

ELIGIBILITY:
Patient Selection and Data Collection This study will be implemented in a single institution, Diyarbakır Gazi Yaşargil Training and Research Hospital, which functions as a tertiary cancer treatment facility.

Between March 2025 and December 2025, patients with newly diagnosed clinical early stage (FIGO 2023 stages 1 and 2) endometrial cancer who will be treated with laparoscopic surgical staging with SLN mapping at our institution will be randomized into groups. The research procedure has been approved by the ethics committee/institutional review board of Diyarbakır Gazi Yaşargil Training and Research Hospital and informed consent signed by the patient will be included in each table reviewed.

Eligible participants will be required to give informed consent to participate in the study.

Inclusion criteria will include

* Participants whose endometrial biopsy resulted in endometrial cancer and whose disease will be detected limited to the uterus using imaging modalities (computed tomography [CT], magnetic resonance imaging or Fluorine-18 fluorodeoxyglucose positron emission tomography/CT)
* Absence of synchronous malignancies.
* No neoadjuvant treatment before surgical intervention.

Exclusion criteria will include:

* Contraindications to using methylene blue dye or contraindications to the vNOTES procedure.
* Patients who have had previous malignancy surgery.
* Severe, deeply penetrating endometriosis or enlarged uterus that may require forced vaginal extraction
* Receiving neodajuvant therapy

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Total operation duration | During surgery
  The total duration of the operation in minutes
Duration of right and left lymphadenectomy | During surgery
  The duration of lymphadenectomies in minutes
Number of lymph nodes excised | Postoperative second week
  Lymph node count in the pathology report
number of positive lymph nodes | Postoperative second week
  Sentinel positive lymph nodes in the pathology report
Hospitalization duration | During hospital stay
  Number of days patients stayed at the hospital postoperatively
Total bleeding volume | During surgery
  Measured by the suction bottle's volume and number of surgical gauzse used during surgery
Difference between pre- and postoperative hemoglobin values | Postoperative 1st day
  Hemoglobin level (g/dL)
Surgical complications | During hospital stay
  Clavien dindo scale of surgical complications
Location o SLN | During surgery
  The area that sentinel lymph node detected internal iliac, external iliac ,bifurcation or obturator fossa
Preoperative and postoperative hematocrit values | During hospital stay
  Hematocrit level (%)
Tumor's patological features | Postoperative second week
  Histophatology, grade, lymphovascular invasion, tumor diameter(cm), myometrial invasion, stage, total positive lymph node count
Management of complications | through study completion
  intraoperative and postoperative complication's management
Duration of lateral colpotomy | During surgery
  at transvaginal retroperitoneal procedure ; before the lymphadenectomy we are making and incision to the lateral of cervix .this time describes the time that to reach the obturator fossa to pick the nodes.
Duration of hysterectomy | During surgery
  minutes
Sentinel lymphnode's side and number | Postoperative second week
  number

SECONDARY OUTCOMES:
Postoperative pain | 3rd and 6th month after operation
  visual analogue scale, higher scores indicate worse pain
Sexual function | at postoperative 3rd and 6th month
  assessed by Female Sexual Function Index, higher scores indicate greater satisfaction
Timing of passing gas | During hospital stay
  Bowel function
Demographic features | Postoperative second week
  Age, gravidity, parity, previous vaginal delivery, body-mass index
Previous abdominal surgery | Preoperative day
  Medical history
Initiation of mobilization | During hospital stay
  After operation the time (hour) that paient is avaliable to mobilize out from the bed
6th hour and 24th hour VAS score | postoperatively 6th and 24th hours score
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

CONTACTS AND LOCATIONS:
Overall Officials: Behzat Can, Assoc. Prof., Study Chair — Health Sciences University Gazi Yasargil Training and Research Hospital; Sedat Akgol, Assoc. Prof., Study Director — Health Sciences University Gazi Yasargil Training and Research Hospital; Kevser Arkan, MD, Principal Investigator — Health Sciences University Gazi Yasargil Training and Research Hospital
Locations (1):
- Gazi Yasargil Training And Research Hospital, Diyarbakır, Baglar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: It will be shared when the study is published.
Access Criteria: When the study is published, the data will be shared by the corresponding author on request.

REFERENCES:
- [Background] Deng L, Liu Y, Yao Y, Deng Y, Tang S, Sun L, Wang Y. Efficacy of vaginal natural orifice transluminal endoscopic sentinel lymph node biopsy for endometrial cancer: a prospective multicenter cohort study. Int J Surg. 2023 Oct 1;109(10):2996-3002. doi: 10.1097/JS9.0000000000000551. PMID 37335988
- [Background] Can B, Akgol S, Adiguzel O, Kaya C. A new, less invasive approach for retroperitoneal pelvic and para-aortic lymphadenectomy combining the transvaginal natural orifice transluminal endoscopic surgery (vNOTES) technique and single-port laparoscopy. Int J Gynecol Cancer. 2024 May 6;34(5):789-790. doi: 10.1136/ijgc-2023-005093. No abstract available. PMID 38316443
- [Background] Baekelandt J, Jespers A, Huber D, Badiglian-Filho L, Stuart A, Chuang L, Ali O, Burnett A. vNOTES retroperitoneal sentinel lymph node dissection for endometrial cancer staging: First multicenter, prospective case series. Acta Obstet Gynecol Scand. 2024 Jul;103(7):1311-1317. doi: 10.1111/aogs.14843. Epub 2024 Apr 16. PMID 38623778